CLINICAL TRIAL: NCT07341893
Title: Clinical Study Evaluating Efficacy and Safety Sacubitril-valsartan in Patients With Heart Failure.
Brief Title: Sacubitril-valsartan in Patients With Heart Failure.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sacubitril-valsartan
Record Dates: First submitted 2026-01-01; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: NT-proBNP; Galectin 3; GDF-15; Sacubitril -Valsartan
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Adrenergic beta-Antagonists

STUDY DESIGN:
Intervention Model Description: 60 patients with heart failure reduced ejection fraction, patients, will be consecutively randomized into two groups, the first group (n=30) will be given Sacubitril-valsartan twice daily and the second group (n=30) on standard treatment of heart failure.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacubitril-valsartan group (Active Comparator): group (n=30) will be given Sacubitril-valsartan twice daily plus standard treatment.
  Interventions: Drug: Sacubitril-valsartan
- Control group (Placebo Comparator): Control group (n=30) on standard treatment of heart failure.
  Interventions: Drug: standard treatment of heart failure

INTERVENTIONS:
Drug: Sacubitril-valsartan — patients (n=30) will be given Sacubitril-valsartan 50 mg twice daily.
  Other Names: Entresto
  Arms: Sacubitril-valsartan group
Drug: standard treatment of heart failure — Control group (n=30) on standard treatment of heart failure.
  Other Names: Beta blockers, ACEis
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of Sacubitril -Valsartan in patients with heart failure.

DETAILED DESCRIPTION:
* A 3-month, prospective interventional study, which will include 60 patients with heart failure reduced ejection fraction, patients, will be consecutively randomized into two groups, the first group (n=30) will be given Sacubitril-valsartan twice daily and the second group (n=30) on standard treatment of heart failure.
* Approval will be obtained from Research and Ethics Committee of Faculty of Pharmacy, Damanhour University. Patients will provided written informed consent and will be checked for inclusion and exclusion criteria.
* All patients will undergo analysis of inflammatory biomarkers such as: NT-proBNP, Galectin-3 and GDF-15 at beginning of the study and after 3 months of the study.
* Echocardiography study before and after the study focusing on:

Measurement of parameters such as: Left atrial diameter (LAD), basic left ventricular dimensions (EDD and ESD), Ejection fraction (EF%).

- Follow up will be performed for assessing:

1. MACE such as MI, stroke, HF, or death.
2. LV Echocardiography improvements of any of basic Echo parameters.
3. Assessment of New York Heart association (NYHA) class.

Outcomes: all patients will be followed up for 3 months for:

* 1ry outcomes: A.Major Adverse Cardiovascular Events (MACE) such as MI, stroke or death. B.Heart failure hospitalization C.LV Echocardiography improvements of any of basic Echo parameters such as: Left atrial diameter (LAD), basic left ventricular dimensions (EDD and ESD), Ejection fraction (EF%).
* 2ry outcomes: Change in inflammatory markers such as: NT-proBNP, GDF-15 and Galectin-3.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old for both genders.
* LV ejection fraction (LVEF) ≤40%.
* Heart failure patients with NYHA grade II-IV.

Exclusion Criteria:

1. CKD with GFR < 20 ml/min/1.73
2. Serum potassium < 5.5 mmol / L.
3. Pregnant or lactating women
4. Active infection.
5. Congenital heart disease.
6. Autoimmune disorders or connective tissue disorders.
7. Severe hepatic dysfunction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
MACE incidence | 3 months
  Major Adverse Cardiovascular Events (MACE) such as MI, stroke or death.
Ejection fraction (EF%) | 3 months
  Ejection fraction (EF%) improvement.

SECONDARY OUTCOMES:
NT-proBNP level (pg/ml) | 3 months
  Change in NT-proBNP level
Galectin-3 level (pg/ml) | 3 months
  Change in Galectin-3 level
GDF-15 level (pg/ml) | 3 months
  Change in GDF-15 level

CONTACTS AND LOCATIONS:
Overall Officials: Nouran A. Abu Shaara, Bachlore, Principal Investigator — Damanhour University
Locations (1):
- Damanhur Medical National Institute, Damanhūr, Elbehairah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu H, Claggett BL, Packer M, Lam CSP, Swedberg K, Rouleau J, Zile MR, Lefkowitz M, Desai AS, Jhund P, McMurray JJV, Solomon SD, Vaduganathan M. Effects of Sacubitril/Valsartan on All-Cause Hospitalizations in Heart Failure: Post Hoc Analysis of the PARADIGM-HF and PARAGON-HF Randomized Clinical Trials. JAMA Cardiol. 2024 Nov 1;9(11):1047-1052. doi: 10.1001/jamacardio.2024.2566. PMID 39210725
- [Background] Lee YH, Lin PL, Chiou WR, Huang JL, Lin WY, Liao CT, Chung FP, Liang HW, Hsu CY, Chang HY. Combination of ivabradine and sacubitril/valsartan in patients with heart failure and reduced ejection fraction. ESC Heart Fail. 2021 Apr;8(2):1204-1215. doi: 10.1002/ehf2.13182. Epub 2021 Jan 6. PMID 33410280